CLINICAL TRIAL: NCT00372515
Title: Phase I Study of High Dose Gefitinib (Iressa) for the Treatment of Carcinomatous Meningitis in Adult Patients With Non-Small Cell Lung Cancer and Known or Suspected EGFR Mutations
Brief Title: High Dose Gefitinib for the Treatment of Carcinomatous Meningitis in Adult Patients With Non-Small Cell Lung Cancer and Known or Suspected EGFR Mutations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David M. Jackman, MD (Other)
Collaborators: AstraZeneca (Industry); Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, David M. Jackman, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-403
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: epidermal growth factor; EGFR; lung cancer; Iressa; Gefitinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High dose gefitinib (Experimental)
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — On days 1-14 gefitinib will be taken orally daily at either 750, 1000, or 1250mg (depends upon when subject entered trial). If medication is tolerated well, subject will take 500mg daily on days 15-28 of each 28-day cycle. Cycles (higher dose followed by lower dose) will be repeated as long as subject's cancer does not worsen and they do not experience any serious side effects.
  Other Names: Iressa

SUMMARY:
The primary purposes of this study are to find out if using high doses of the drug Gefitinib (Iressa) as a way to treat patients with non-small cell lung cancer that has spread to the covering of the brain and/or spinal cord (meninges) results in any bad side effects; and to determine the highest dose that can be given to patients in this setting.

DETAILED DESCRIPTION:
* The standard therapy for this type of cancer is to give chemotherapy directly into the spinal fluid, usually by a spinal tap. Some chemotherapy may, in some cases, be combined with radiation. This study looks at a different way of treating this type of cancer.
* This study is specifically for patients whose lung cancer has changes in a protein called the epidermal growth factor receptor (EGFR). The study drug, gefitinib, was developed to stop the signals from the EGFR that tell certain types of lung cancers tumors to grow. By using higher doses than are normally used, we hope to increase the amount of drug in the spinal fluid to attempt to kill the cancer cells around the spinal cord and brain.
* Since we are looking for the highest dose of gefitinib that can be given safely, not everyone who participates in this study will be receiving the same amount of drug.
* Patients will start taking gefitinib daily by mouth on Day 1 and will continue taking this medication daily at home. On the first day the patient takes gefitinib and on Day 14 of each treatment cycle (1 cycle equals 28 days), the patient will undergo: Physical examination by the study doctor and a detailed neurological exam by a neuro-oncologist; sampling of cerebrospinal fluid (CSF) by lumbar puncture; review of current medications; measurement of vital signs; check on the patients ability to perform daily activities; blood work.
* If the patient is tolerating the study medication well, then the patient will receive a lower dose for days 15-28 of the cycle.
* At the end of each cycle on Day 28, the patient will meet with the study doctor and have the following: a physical examination; review of current medications; measurement of vital signs, check on the patients ability to perform daily activities; blood tests; MRI of the brain and spinal cord to assess tumor response; every two cycles a CT scan of the chest and abdomen to assess the tumor response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of non-small cell lung cancer of any histologic subtype
* High likelihood of gefitinib sensitivity, as evidenced by one or more of the following: previous complete or partial response to treatment with an epidermal growth factor receptor-tyrosine kinase inhibitor, erlotinib, or gefitinib; known somatic mutation of the EGFR tyrosine kinase
* Recurrent or persistent disease as manifested by carcinomatous meningitis
* ECOG PS 0-3
* Age 18 years or older
* Greater than 2 weeks since prior radiation therapy
* Greater than 3 weeks since prior major surgery
* Adequate hematologic, renal, and/or hepatic function
* Coagulation parameters: international normalized ratio(INR)less than or equal to 1.5 and an activated thromboplastin time < 50 seconds

Exclusion Criteria:

* Previous Grade 4 toxicity on gefitinib or erlotinib leading to dose reduction or interruption
* Uncontrolled brain metastases, or brain metastases associated with mass effect that would contraindicate lumbar puncture
* Any other malignancy within the past five years, except for adequately treated carcinoma of the cervix, basal or squamous cell carcinomas of the skin
* Dysphagia
* Active gastrointestinal disease or disorder that alters gastrointestinal motility or absorption
* Incomplete healing from previous oncologic or other major surgery
* Any pre-existing severe or unstable medical condition
* Any condition requiring concurrent and ongoing use of anticoagulation
* Inability to undergo collection of CSF, either by repeated lumbar puncture or placement of an Omaya reservoir
* Pregnant or breastfeeding
* Concurrent intrathecal drug administration or radiotherapy
* Concurrent systemic chemotherapy or investigational agent
* Anticoagulant except aspirin or heparin flushes
* Enzyme-inducing anti-epileptic drug
* CYP3A4 inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-06; Primary Completion 2012-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To assess the safety of administering gefitinib in doses of 750mg to 1250mg in adult patients with carcinomatous meningitis from non-small cell lung cancer with known or suspected somatic EGFR mutations. | 2 years

SECONDARY OUTCOMES:
To measure the cytologic response rate, response duration, time to neurologic progression, and survival following high dose gefitinib therapy administered on this schedule | 2 years
to measure gefitinib levels with serum and cerebrospinal fluid while on therapy, and to correlate these levels with toxicity, response and survival | 2 years
to examine archived tumors for the presence or absence of EGFR mutations and resistance mutations, and to correlate those mutations with cytologic response, time to neurologic progression, and survival. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Johnson, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Jackman DM, Cioffredi LA, Jacobs L, Sharmeen F, Morse LK, Lucca J, Plotkin SR, Marcoux PJ, Rabin MS, Lynch TJ, Johnson BE, Kesari S. A phase I trial of high dose gefitinib for patients with leptomeningeal metastases from non-small cell lung cancer. Oncotarget. 2015 Feb 28;6(6):4527-36. doi: 10.18632/oncotarget.2886. PMID 25784657